CLINICAL TRIAL: NCT00730548
Title: Clinical Evaluation to Assess the Effect of the Combination of a Pre-Defined Management Pathway to Reduce Fluid Overload in Cardiac Decompensation With Carelink Remote Management, Connexus Remote Telemetry and the OptiVol Early Warning System on Health Care Utilization
Brief Title: Compare Remote Patient Management and Standard Care in CRT-D and ICD-patients to Assess the Effect on Heart Failure
Acronym: ConnectOptiVol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEN_G_CA_7
Record Dates: First submitted 2008-06-19; First posted 2008-08-08 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure; Ventricular Tachycardia; Cardiac Desynchronization
MeSH Terms: conditions — Heart Failure; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Remote Arm (OptiVol plus Connexus Telemetry plus CareLink plus Intervention Algorithm), Clinical Management Alerts ON
  Interventions: Behavioral: Device triggered remote telephone contact because of Care Alert
- 2 (No Intervention): No Care Alerts available, standard treatment of the patient

INTERVENTIONS:
Behavioral: Device triggered remote telephone contact because of Care Alert — Care Alerts on, physician will be notified in case of an Care Alert. Depending on the outcome of the telephone contact drug adjustment and / or further interventions can be prescribed
  Other Names: OptiVol; CareLink; Medtronic Concerto; Medtronic Consulta; Medtronic Secura; Medtronic Virtuoso
  Arms: 1

SUMMARY:
This pilot study is to prospectively evaluate the benefit of clinicians being able to access ICD device information in a timelier manner and treat fluid overload with a pre-defined pattern using the Medtronic OptiVol, Medtronic CareAlerts and Medtronic CareLink in Conexus-enabled devices (remote arm) as compared to the same devices without Medtronic OptiVol, Medtronic CareAlerts and Medtronic CareLink available to the treating physician (standard arm).

ELIGIBILITY:
Inclusion Criteria:

* Implantation of a market-approved Medtronic Connexus CRT-D- or DR-ICD-device
* Patient consents to study
* Ability to replace follow-ups with CareLink follow-ups
* Ability to attend all follow-ups at study center

Exclusion Criteria:

* Permanent AF
* Less than 18 years of age
* Life expectancy less than 15 months
* Participation in another clinical study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-11; Primary Completion 2011-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Time to first hospitalization due to worsened heart failure | 15 months

SECONDARY OUTCOMES:
Time from device detected onset of arrhythmias, cardiovascular disease progression and system issues to clinical decision making | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zabel, MD, Principal Investigator — University Hospital of Goettingen
Locations (1):
- University Hospital of Goettingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zabel M, Vollmann D, Luthje L, Seegers J, Sohns C, Zenker D, Hasenfuss G. Randomized Clinical evaluatiON of wireless fluid monitoriNg and rEmote ICD managemenT using OptiVol alert-based predefined management to reduce cardiac decompensation and health care utilization: the CONNECT-OptiVol study. Contemp Clin Trials. 2013 Jan;34(1):109-16. doi: 10.1016/j.cct.2012.10.001. Epub 2012 Oct 13. PMID 23073567
- [Result] Luthje L, Vollmann D, Seegers J, Sohns C, Hasenfuss G, Zabel M. A randomized study of remote monitoring and fluid monitoring for the management of patients with implanted cardiac arrhythmia devices. Europace. 2015 Aug;17(8):1276-81. doi: 10.1093/europace/euv039. Epub 2015 May 17. PMID 25983310